CLINICAL TRIAL: NCT05655949
Title: A Single Arm Phase 2 Study of Y-90 SIRT in Combination With Durvalumab (MEDI 4736) and Gemcitabine/Cisplatin in Locally Advanced, Unresectable or Metastatic Intrahepatic Cholangiocarcinoma
Brief Title: Y-90 With Durvalumab/Gem/Cis in Intrahepatic Cholangio
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: AstraZeneca (Industry); Sirtex Medical (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Andrea Bullock, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-541
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Bile Duct Cancer; Cholangiocarcinoma; Cholangiocarcinoma Non-resectable; Cholangiocarcinoma Metastatic; Metastatic Intrahepatic Cholangiocarcinoma
Keywords: Bile Duct Cancer; Cholangiocarcinoma; Cholangiocarcinoma Non-resectable; Cholangiocarcinoma Metastatic; Metastatic Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Bile Duct Neoplasms; Cholangiocarcinoma | interventions — Gemcitabine; Cisplatin; durvalumab; Yttrium-90

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Gemcitabine + Cisplatin + Durvalumab + Yttrium-90 Selective Internal Radiation Therapy (Experimental): Participants will receive:
  * Cycle 1:
  Day 1 of 21 Day cycle: Pre-determined dose(s) of Gemcitabine and Cisplatin (Chemotherapy) plus Durvalumab (immunotherapy).
  Day 8 of 21 Day cycle: Pre-determined dose(s) of Gemcitabine and Cisplatin (Chemotherapy)
  Week 2 or 3 of 21 Day Cycle: One time treatment of Y-90 radiation.
  * Cycles 2-8:
  Day 1 of 21 Day cycle: Pre-determined dose(s) of Gemcitabine and Cisplatin (Chemotherapy) plus Durvalumab (immunotherapy).
  Day 8 of 21 Day cycle: Pre-determined dose(s) of Gemcitabine and Cisplatin (Chemotherapy)
  * Cycles 9+:
  Day 1 of 21 Day Cycle: Durvalumab (immunotherapy) maintenance
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Durvalumab; Radiation: Yttrium-90

INTERVENTIONS:
Drug: Gemcitabine — Intravenous infusion
  Other Names: Gemzar
Drug: Cisplatin — Intravenous infusion
  Other Names: Platinol; Platinol®-AQ
Drug: Durvalumab — Intravenous infusion
  Other Names: Imfinzi
Radiation: Yttrium-90 — Injection of radiation microsphere beads

SUMMARY:
This trial is designed to study a combination of interventions (chemotherapy, immunotherapy, and radiation) as a potential new treatment for bile duct cancer that cannot be removed with surgery.

The specific names of the interventions that will be used are:

* Y-90 (a type of radiation microsphere bead)
* Durvalumab (a type of immunotherapy)
* Gemcitabine (a type of chemotherapy)
* Cisplatin (a type of chemotherapy)

DETAILED DESCRIPTION:
This is a single arm Phase II, non-randomized, open-label clinical trial assessing the safety and efficacy of Y-90 SIRT in combination with durvalumab, gemcitabine and cisplatin in participants with locally advanced unresectable or metastatic intrahepatic cholangiocarcinoma.

The U.S. Food and Drug Administration (FDA) has approved durvalumab for bile duct cancer that cannot be removed with surgery, but it has been approved for other uses.

The U.S. Food and Drug Administration (FDA) has already approved gemcitabine, cisplatin, and Y-90 microsphere radiation as a treatment option for bile duct cancer that cannot be removed with surgery.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits. Participants will be followed for up to 52 weeks if taken off protocol therapy.

It is expected that about 30 people will take part in this research study.

AstraZeneca, a pharmaceutical company, is supporting this research study by providing one of the study drugs, durvalumab, as well as providing research funding.

Sirtex, a medical device company, is supporting this research by providing the Y-90 radiation microsphere beads.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study
* Male and female participants at least 18 years of age at the time of signing the ICF
* Histologically or cytologically confirmed locally advanced unresectable or metastatic intrahepatic cholangiocarcinoma; at least one intrahepatic lesion must be present
* Radiographically measurable or evaluable disease by CT or MRI per RECIST v1.1 criteria
* ECOG performance status ≤1
* Body weight >30 kg
* Must have a life expectancy of at least 12 weeks
* Participants must have adequate marrow function as defined below:

  * Hemoglobin ≥9.0 g/dL
  * Absolute neutrophil count (ANC) ≥1.0 × 109 /L
  * Platelet count ≥75 × 109/L
* Participants must have adequate renal function as defined below:

  * Serum creatinine ≤ 1.5 mg/dL OR
  * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
* Participants must have adequate hepatic function as defined below:

  * Bilirubin ≤1.5 x ULN
  * ALT ≤ 2.5 x ULN unless liver metastases are present, in which case it must be ≤5x ULN
  * AST ≤ 2.5 x ULN unless liver metastases are present, in which case it must be ≤5x ULN
  * This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician
  * No known history of active HBV or HCV infection.

    * Note: Participants with Hepatitis C who have been clinically cured, defined as persistent absence of Hepatitis C RNA detected by polymerase chain reaction (PCR) test in serum 12 weeks after completing antiviral treatment, are eligible for this study
    * Note: Participants with a history of Hepatitis B infection that are currently on viral suppressive therapy are eligible for enrollment
* Adequate coagulation studies as demonstrated by prothrombin (PT) and partial thromboplastin (PTT) time within normal limits (</= 1.5 x ULN) in the absence of anticoagulation medication. Participants receiving anticoagulation may be approved by sponsor
* Participants with known human immunodeficiency virus (HIV) on effective highly-active antiretroviral therapy (HAART) with undetectable viral load within 6 months are eligible for this trial, so long as the following criteria are met:

  * HAART does not interact with or have overlapping toxicities with study medication, per discretion of the treating provider
  * CD4 count is ≥350 cells/uL, viral load is undetectable, and not taking prohibited cytochrome (CYP)-interacting medications
  * Probable long-term survival with HIV if cancer were not present
  * Stable on a HAART regimen for ≥4 weeks and willing to adhere to their HAART regimen with minimal overlapping toxicity and drug-drug interactions with the experimental agents in this study
  * HIV is not multi-drug resistant
  * Taking medication and/or receiving antiretroviral therapy that does not interact or have overlapping toxicities with the study medication

Exclusion Criteria:

* Surgically resectable disease at enrollment
* Histologically or cytologically confirmed diagnosis of primary hepatocellular carcinoma or mixed adenocarcinoma/hepatocellular carcinoma
* Received prior systemic chemotherapy and/or radiotherapy for intrahepatic cholangiocarcinoma. Prior surgical resection and adjuvant chemotherapy or chemoradiotherapy is allowed if more than 6 months have elapsed since last dose of treatment, and if the tumor is amenable to Y-90 SIRT
* Prior treatment with anti-PD-1, anti-PD-L, including durvalumab antibody, or any other drug treatment specifically targeting T-cell co-stimulation or checkpoint pathways
* Any of the following within 6 months of screening:

  * New York Heart Association (NYHA) Class III or IV heart failure
  * Myocardial infarction, unstable angina pectoris, or symptomatic coronary artery disease
  * Unstable arrhythmia
  * Stroke to transient ischemic attack
* Previous malignancies, except for adequately treated non-melanoma skin cancer, in-situ cancer, or any other cancer from which the subject has been disease-free for at least 3 years
* Severe chronic obstructive or other pulmonary disease with chronic baseline hypoxemia due to potential for gemcitabine-induced bronchospasm and/or durvalumab-induced pneumonitis
* Major surgery (other than diagnostic) within 4 weeks of study treatment day 1
* Active, uncontrolled or untreated bacterial, viral, or fungal infection that requires systemic therapy
* Active, untreated HIV, HBV, or HCV
* Subjects who have participated in another investigational drug or device study within 4 weeks prior to study registration.

Pregnant women are excluded from this study because cisplatin is a class D agent with the potential for teratogenic or abortifacient effects. Because cisplatin is present in breast milk and there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cisplatin, breastfeeding should be discontinued prior to entry into the study. Subjects and their sexual partners entered into the study must agree to contraception. The following restrictions apply while the patient is receiving study treatment and for the specified times before and after:

* Female patients of child-bearing potential Female patients of childbearing potential who are not abstinent and intend to be sexually active with a non sterilized male partner must use at least 1 highly effective method of contraception (Table 2) from the time of screening throughout the total duration of the drug treatment and the drug washout period (90 days after the last dose of durvalumab monotherapy). Non-sterilised male partners of a female patient of childbearing potential must use male condom plus spermicide throughout this period. Cessation of birth control after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Female patients should also refrain from breastfeeding throughout this period.
* Male patients with a female partner of childbearing potential Non-sterilized male patients who are not abstinent and intend to be sexually active with a female partner of childbearing potential must use a male condom plus spermicide from the time of screening throughout the total duration of the drug treatment and the drug washout period (90 days after the last dose of durvalumab monotherapy). However, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Male patients should refrain from sperm donation throughout this period.

Female partners (of childbearing potential) of male patients must also use a highly effective method of contraception throughout this period (Table 2).

Females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal.

Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

* Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution.
* Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago.

Highly effective methods of contraception, defined as one that results in a low failure rate (ie, less than 1% per year) when used consistently and correctly are described in Table 2. Note that some contraception methods are not considered highly effective (e.g. male or female condom with or without spermicide; female cap, diaphragm, or sponge with or without spermicide; non-copper containing intrauterine device; progestogen-only oral hormonal contraceptive pills where inhibition of ovulation is not the primary mode of action [excluding Cerazette/desogestrel which is considered highly effective]; and triphasic combined oral contraceptive pills).

* Copper T intrauterine device
* Levonorgestrel-releasing intrauterine system (e.g., Mirena®)a
* Implants: Etonogestrel-releasing implants: e.g. Implanon® or Norplant®
* Intravaginal: Ethinylestradiol/etonogestrel-releasing intravaginal devices: e.g. NuvaRing®
* Injection: Medroxyprogesterone injection: e.g. Depo-Provera®
* Combined Pill: Normal and low dose combined oral contraceptive pill
* Patch: Norelgestromin/ethinylestradiol-releasing transdermal system: e.g. Ortho Evra® Minipillc: Progesterone based oral contraceptive pill using desogestrel: Cerazette® is currently the only highly effective progesterone-based

  * Any concomitant disease or condition that could interfere with the conduct of the study, or that would in the option of the investigator pose an unacceptable risk to the subject in the study
  * Contraindications to Y-90 SIRT per assessment by treating Interventional Radiologist (eg significant vascular drainage of the tumor to the lung that increases the potential for pulmonary toxicity)
  * Unwillingness or inability to comply with the study protocol
  * History of allogenic organ transplantation.
  * Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
  * Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
  * History of active primary immunodeficiency
  * Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice
  * Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
  * Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
  * Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
  * Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Median Progression Free Survival (PFS) | Enrollment to end of treatment and up to 52 weeks thereafter
  PFS is defined as the time from date of entry into the study until the date of disease progression (according to RECIST v1.1 and assessed by an independent central reviewer) or death, whichever occurs first.
Incidence of Grade 3 or Higher Treatment-Related Toxicity | Enrollment to end of treatment and up to 52 weeks thereafter
  All grade 3 or higher adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 as reported on case report forms. Incidence is the number of patients experiencing at least one treatment-related grade 3 or higher AE of any type during the time of observation.

SECONDARY OUTCOMES:
Median Overall Survival (OS) | Enrollment to end of treatment and up to 52 weeks thereafter
  OS is based on Kaplan-Meier method and defined as the time from date of entry into the study until the date of death.
Objective Response Rate (ORR) | Enrollment to end of treatment and up to 52 weeks thereafter
  ORR is defined as the proportion of participants with the best overall response of complete response or partial response according to RECIST v1.1 criteria as assessed by an independent central reviewer"
Disease Control Rate (DCR) | Enrollment to end of treatment and up to 52 weeks thereafter
  DCR is defined as the proportion of participants with the best overall response of complete response, partial response, or stable disease according to RECIST v1.1 criteria as assessed by an independent central reviewer

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Bullock, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu